CLINICAL TRIAL: NCT02510729
Title: Sphenopalataine Ganglion (SPG) Stimulation in Cluster Headache Patients
Brief Title: SPG Neurostimulation in Cluster Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-15005609
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPG neurostimulation (Active Comparator): Sphenopalatine ganglion (SPG) neurostimulation of 20 Hz
  Interventions: Device: Neurostimulation
- Sham Stimulation (Placebo Comparator): Sham stimulation with amplitude=0
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Neurostimulation
  Arms: SPG neurostimulation
Device: Sham stimulation
  Arms: Sham Stimulation

SUMMARY:
We hypothesized that LF stimulation of the SPG would increase parasympathetic outflow, activate sensory afferents and provoke a cluster-like attack.

DETAILED DESCRIPTION:
We conducted a double-blind, randomized, sham-controlled, crossover study to investigate cluster attack induction following LF (20 Hz and 0.2-2.1 amplitude) and sham (amplitude = 0) stimulation in 20 CH patients with implanted SPG neurostimulator. In addition, we measured plasma concentrations of pituitary adenylate cyclase-activating polypeptide-38 (PACAP38) and vasoactive intestinal peptide (VIP), as markers for parasympathetic activation before, during and after SPG stimulation. We also investigated if LF SPG stimulation induces changes in cardiac autonomic regulation and whether any attacks induced by SPG stimulation are associated with such changes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cluster patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of cluster-like attacks and cephalic autonomic symptoms | 0-60 min
  Difference in incidence of cluster-like attacks and cephalic autonomic symptoms between LF and sham stimulation.

SECONDARY OUTCOMES:
Mechanical detection and pain thresholds | 0-60 min
  Difference in mechanical detection and pain thresholds in the face between LF and sham stimulation measured by pin-prick and von Frey hairs.
Plasma concentrations of PACAP38 and VIP | 0-60 min
  Difference in plasma concentrations of PACAP38 and VIP between LF and sham stimulation.
Cardiac autonomic regulation (HRV) | 0-60 min
  Changes in cardiac autonomic regulation (HRV) between LF and sham stimulation and during cluster attacks measured by continious ECG.
Mean arterial blood pressure and heart rate | 0-60 min
  Difference in mean arterial blood pressure and heart rate between LF and sham stimulation.
Headache intensity | 0-60 min
  Difference in headache intensity measured by numerical rating scale (NRS 0-10) between LF and sham stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Prof., Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Guo S, Petersen AS, Schytz HW, Barlose M, Caparso A, Fahrenkrug J, Jensen RH, Ashina M. Cranial parasympathetic activation induces autonomic symptoms but no cluster headache attacks. Cephalalgia. 2018 Jul;38(8):1418-1428. doi: 10.1177/0333102417738250. Epub 2017 Oct 30. PMID 29082824